CLINICAL TRIAL: NCT05878015
Title: A Randomized Study Comparing Intravenous (IV) Acetaminophen to Usual Care for Pain Management for Small Bowel Obstruction - Feasibility Study
Brief Title: A Study of Intravenous Acetaminophen for Small Bowel Obstruction
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tatjana Gavrancic, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-000547
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Small Bowel Obstruction
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV Acetaminophen Group (Experimental): Subjects presented to emergency department (ED) and diagnosed with small bowel obstruction which receive IV acetaminophen
  Interventions: Drug: Acetaminophen
- Usual Care Group (No Intervention): Subjects presented to emergency department (ED) and diagnosed with small bowel obstruction will receive intravenous opioids per their provider's choice as standard of care.

INTERVENTIONS:
Drug: Acetaminophen — 1000mg intravenous every 6 hours on day 1 and day 2. 1000mg intravenous every 8 hours on day 3 as needed.
  Other Names: Tylenol
  Arms: IV Acetaminophen Group

SUMMARY:
The purpose of this study is to compare IV Acetaminophen for pain control to the usual care with opioids in patients admitted for small bowel obstruction.

DETAILED DESCRIPTION:
The primary aim of this study is to assess the feasibility of conducting a randomized trial involving intravenous acetaminophen for pain control compared to usual care with opioids in patients admitted for small bowel obstruction and to summarize pain scores up to 72 hours after treatment. Patients presented and diagnosed with small bowel obstruction (SBO) will be screened for eligibility and will be offered participation in this study. Patients admitted for SBO for medical management with pain on admission will be eligible to participate in study. This will include patients with malignant and nonmalignant SBO. Participants will be randomly assigned into one of two groups, either the Treatment Group which receive IV acetaminophen or the Usual Care Group which will receive intravenous morphine or hydromorphone as needed for pain control. A Nasogastric (NG) tube will be placed when it is indicated, if patient is having significant nausea or vomiting. Pain scores will be followed as usual pain management assessment and reported in the medical record. Once SBO is resolved (usually 3 days after admission), active study participation will end. Participants may be followed via their medical record up to 30 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Small bowel obstruction diagnosed by radiographic study; and
* Abdominal pain on admission.
* Nothing per mouth diet.
* The ability to give appropriate consent or have an appropriate representative available to do so.

Exclusion Criteria:

* Known liver failure or cirrhosis.
* Acetaminophen toxicity on admission.
* Known acetaminophen allergy.
* Alcohol intoxication on admission.
* History of substance abuse.
* Creatinine clearance < 30 (or Creatinine level > 2).
* Liver transplant recipients.
* Ileus on admission.
* Admitted for surgical intervention for SBO.
* Admitted for venting Gastric tube placement.
* On chronic opioid therapy (defined as use of opioid on daily or near daily basis within previous 45 days (both long acting and short acting).
* Presentation without abdominal pain on admission.
* Already hospitalized for other reasons and develop SBO while at the hospital.
* Pregnant women.
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Resolution of small bowel obstruction | 3 days
  Days until small bowel obstruction resolution, measured by admission date to date that diet was placed
Pain Scores | 3 days
  Pain is measured by a pain scale of subjective pain reported by patients and measured by nurses and ranges from 0 (no pain) to 10 (worst pain).
Length of hospital stay | 3 days
  Measured by days from admission day to discharge day

SECONDARY OUTCOMES:
Death | 3 days
  Number of subject deaths
Bowel Perforation | 3 days
  Number of subject to experience a bowel perforation
Surgery | 3 days
  Number of subjects to require surgical intervention for small bowel obstruction treatment
Allergic reaction to acetaminophen | 3 days
  Number of subjects to experience an allergic reaction to acetaminophen

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Gavrancic, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of Intravenous Acetaminophen for Small Bowel Obstruction — https://www.mayo.edu/research/clinical-trials/cls-20548880